CLINICAL TRIAL: NCT03940105
Title: The Effects of Snack Size and Variety on Appetite Control, Satiety, and Eating Behavior in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Sabra Dipping Company, LLC (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1807020783
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Snacking
Keywords: intuitive eating; package size; food variety

STUDY DESIGN:
Intervention Model Description: tightly-controlled, randomized cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): For 3 days during the control snack pattern, the participants will be asked to complete dietary recalls concerning their afternoon and evening snacking behavior. The participants will use the Automated Self-Administered 24-hour Recall (ASA24) system which was developed by the National Cancer Institute.
- Standard Packout (Active Comparator): This packout contains a variety of foods to be consumed, ad libitum, throughout the remainder of the day following the standardized lunch.
  Interventions: Behavioral: Packout
- Large Package Packout (Active Comparator): This packout contains a variety of foods to be consumed, ad libitum, throughout the remainder of the day following the standardized lunch. It differs from the Standard Packout in that the package sizes of all the foods are larger (though food amount remains the same).
  Interventions: Behavioral: Packout
- Variety Packout (Active Comparator): This packout contains a variety of foods to be consumed, ad libitum, throughout the remainder of the day following the standardized lunch. It differs from the Standard Packout in that there is about twice as much snack variety (though food amount remains the same).
  Interventions: Behavioral: Packout

INTERVENTIONS:
Behavioral: Packout — Each packout provided during 3 of the 4 snack patterns will contain a variety of foods to be consumed, ad libitum, throughout the remainder of the day following the standardized lunch. There are 3 different packouts that will be provided for 3 nonconsecutive weekdays (for a total of 9 packouts). Each packout contains the same calories and types of foods. However, they differ in packaging size and variety.
  Arms: Large Package Packout; Standard Packout; Variety Packout

SUMMARY:
The investigators propose a randomized snack study in normal to obese adults that will test whether snack size, choice, or variety has an influence on daily snack intake.

Aim 1: To validate the in-house packout methodology with 3-day dietary recalls. Aim 2: To examine whether snack variety or snack package size will influence free-living snacking behavior.

Aim 3: To identify whether a correlation exists between mindful eating and free-living snacking behavior.

DETAILED DESCRIPTION:
Participants will complete 4 different snack patterns. Each pattern will include 3 nonconsecutive weekdays (i.e., Monday/Wednesday/Friday; Tuesday/Thursday/Monday, etc.). The snack patterns will be performed at home/work.

The first pattern will simply be a measurement of typical snack habits. For each of the 3 days, the participant will enter all foods and beverages consumed using the online program, Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA-24).

For the other 3 patterns, different snack packouts will be provided to the participant for 3 nonconsecutive weekdays/pattern. The only difference between the packouts is the type of foods provided. The packouts contain commercially available foods commonly eaten by people who snack. Following lunch, the participant will be permitted to eat as much or as little as he/she chooses from the packout until going to bed. Beverages will not be provided and the participant could drink whatever he/she typically consumes.

For all patterns, the participant will be provided with a standardized breakfast, lunch, and dinner to consume at home/work for each of the 3 days/pattern.

ELIGIBILITY:
Inclusion Criteria:

1. age range 18-55 y
2. normal weight to overweight/obese (BMI: 18-32 kg/m2)
3. healthy, non-diabetic
4. not currently or previously on a weight loss or other special diet (in the past 6 months)
5. non-smoking (for the past 6 months)
6. not been clinically diagnosed with an eating disorder
7. habitually eat afternoon/evening snacks at least 4 days/week

Exclusion Criteria:

1. Clinically diagnosed with an eating disorder
2. Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
3. Currently or previously on a weight loss or other special diet (in the past 6 months)
4. Gained/lost >10 lb. over the past 6 months
5. Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 3 months)
6. Not willing or able to complete all study testing procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Ad libitum Snack Energy Intake | 12 testing days across ~4-6 weeks
  Free-living energy intake will be assessed on the three testing days of each testing arm. For the control testing days, the participant will be provided with a standardized breakfast, lunch, and dinner, and will be required to log any snacks consumed on the Automated Self-Administered Recall System (ASA24). For each pack-out testing day, the participant will be provided a standardized breakfast, lunch, and dinner, as well as an excess of snacks to consume, ad libitum, throughout the day. All food items will be initially weighed and recorded. The participants will be instructed to return all uneaten foods as well as all wrappers and containers from consumed food. Any partially eaten, returned items will be weighed accordingly. The snacking and daily energy intake (as well as protein, carbohydrate, sugar, fiber, and fat intake) will be assessed from these pack-outs.
Ad libitum Food Category Intake | 9 testing days across ~3-5 weeks
  Free-living food category intake will be assessed on the three testing days of each packout. The participant will be provided a standardized breakfast, lunch, and dinner, as well as an excess of snacks to consume, ad libitum, throughout the day. All food items will be initially weighed and recorded. The participants will be instructed to return all uneaten foods as well as all wrappers and containers from consumed food. Any partially eaten, returned items will be weighed accordingly. The snack intake of different food categories (i.e. desserts and candy, salty, high fat, high sugar, fruits and vegetables) will be assessed from these pack-outs.

SECONDARY OUTCOMES:
Intuitive Eating Score (1-5) | Baseline (at beginning of study)
  Participant will complete Intuitive Eating Scale-2 survey in order to receive an Intuitive Eating Score. The survey includes a 1 to 5 likert scale with 1 being 'strongly disagree' and 5 being 'strongly agree'. Min score is 1; Max score is 5. The higher the number, the greater the intuitive eating.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Leidy, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in snacking behavior. Data shared will be coded, with no protected health information or identifiable data. A material transfer agreement is requested with approval of the sharing of data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After 6 months following the publication of the study data, data requests can be submitted for approval. The data will be available for up to 24 months post-publication.
Access Criteria: Access can be requested by qualified researchers engaging in independent scientific research. For more information or to submit a request, please contact Heather Leidy at Heather.Leidy@austin.utexas.edu.

REFERENCES:
- [Derived] Reister EJ, Leidy HJ. Snack Package Size and Variety Differentially Influence Energy Intake and Food Choices in Healthy Adults. Curr Dev Nutr. 2022 Jan 17;6(2):nzac004. doi: 10.1093/cdn/nzac004. eCollection 2022 Feb. PMID 35155984